CLINICAL TRIAL: NCT01186900
Title: Comparison of Ultrasound-Guided Needle Aspiration and Open Incision and Drainage in the Management of Cutaneous Abscesses
Brief Title: Comparison of Ultrasound-Guided Needle Aspiration and Open Incision and Drainage for Cutaneous Abscesses
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Dr. Jeffrey Perry, Department of Emergency Medicine, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008198-01H
Record Dates: First submitted 2010-08-19; First posted 2010-08-23 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2011-08

CONDITIONS: Abscess
Keywords: skin abscess; needle aspiration; incision and drainage
MeSH Terms: conditions — Abscess; Surgical Wound | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound-guided needle aspiration (Experimental): One arm is ultrasound-guided needle aspiration, the other active comparison is traditional open incision and drainage of skin abscess
  Interventions: Procedure: ultrasound-guided needle aspiration
- open incision and drainage (Active Comparator)
  Interventions: Procedure: ultrasound-guided needle aspiration

INTERVENTIONS:
Procedure: ultrasound-guided needle aspiration — one time drainage at time of randomization

SUMMARY:
The investigators propose to conduct a, two armed, randomized, controlled pilot study to assess the clinical effects of a) open incision, drainage with daily packing changes, compared to b) Ultrasound guided needle aspiration, in drainage of uncomplicated cutaneous abscesses below the skin surface of adult emergency department patients using concealed allocation in evaluating patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

Patients presenting to the Civic Campus emergency department of The Ottawa Hospital with an abscess less than 5 cm diameter, as judged by the attending emergency physician (measurement with tape measure for diameter) between the hours of 7 am and 10 pm will be approached for possible enrollment. Ultrasound will be used to assess the appropriate exclusion criteria.

Exclusion Criteria:

* Patients under the age of 18 years,
* Patients with a Glasgow coma scale score of <15 (i.e. not completely alert and oriented),
* Patients suspected of having necrotising fascitis,
* Patients with hemodynamic instability (defined as SBP <90, and/or HR >110),
* Patients admitted to hospital,
* Patients who are neither French nor English speaking,
* Patients who are not available for telephone follow-up (i.e. homeless).
* Ultrasound image demonstrates that the abscess is not compressible (generally indicates that the contents of the cyst includes solids, which would not be amenable to aspiration)
* Ultrasound demonstrates that there is no abscess to manage,
* Patients with perianal abscesses who have either Crohn's disease or ulcerative colitis or known perirectal fistula,
* Patients with recurrent abscesses in the same location or abscesses present for more than 2 weeks
* Patients with complex abscesses including deep tissue, sensitive body part involvement which includes: ears, eyes, lacrimal, orbital, submandibular, mouth, peritonsillar, and Bartholin's gland.
* Patients with renal impairment, diabetes, immunocompromised (as these patients are at risk of becoming more ill if an abscess were able to grow).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-06; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction | 7 days

SECONDARY OUTCOMES:
Failure rate | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Woo, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada